CLINICAL TRIAL: NCT00534079
Title: Nasal Inhalation of Dornase Alfa (Pulmozyme) in Patients With Cystic Fibrosis and Chronic Rhinosinusitis - a Double Blind Placebo-controlled Cross-over, Bicenter, Prospective Clinical Study
Brief Title: Nasal Inhalation of Pulmozyme in Patients With Cystic Fibrosis and Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, Head of CF Center, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pulmozyme-nasal-cf
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis; Rhinosinusitis
Keywords: Cystic Fibrosis and chronic rhinosinusitis
MeSH Terms: conditions — Cystic Fibrosis; Rhinosinusitis | interventions — dornase alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dornase alfa (Experimental): 28 days of sinonasal inhalation (Pari Sinus)
  Interventions: Drug: Dornase alfa (Pulmozyme); Drug: isotonic saline
- isotonic saline (Placebo Comparator): 28 days of sinonasal inhalation (Pari Sinus)
  Interventions: Drug: Dornase alfa (Pulmozyme); Drug: isotonic saline

INTERVENTIONS:
Drug: Dornase alfa (Pulmozyme) — 1 x 2,5 ml per day, inhalation use, for 28 days
Drug: isotonic saline — 1 x 2,5 ml per day, inhalation use, for 28 days

SUMMARY:
Rhinosinusitis disorders are often associated with Cystic Fibrosis. They can restrict quality of life enormously and give cause to repeated ENT surgery. The basic defect in CF is a dysfunction of chloride channels in exocrine glands, leading to retention of secretions and consecutive chronic inflammation with bacterial superinfections.

The prospective placebo controlled cross-over study aims at the evaluation of a nasally inhalation of Pulmozyme with respect to mucus retention and resulting inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of cystic fibrosis based on: 3 positive sweat chloride tests and/or genetic characterisation
* Subject is 5 years of age or older
* Subject has chronic or recurrent rhinosinusitic disorders
* Subject is able to comply with the procedures scheduled in the protocol
* Women of childbearing potential are only included into the study, if they are using an effective method of birth control during the protocol (e.g. implants, combined oral contraceptives, injectables, some IUDs, sexual abstinence or vasectomised partner)

Exclusion Criteria:

* Subject has a critical condition defined as: FEV1 < 30% and / or SaO2 < 93% without O2-substitution; need of O2-substitution
* Subject had an ENT surgery within 6 months prior to study
* Subject shows signs of nasal bleeding
* Subject has an ear drum perforation
* Subject had an acute rhinosinusitis or a pulmonary exacerbation at study entry with need of additional systemic antibiotic therapy
* Subject has a new therapy with nasal topic steroids during treatment interval
* Subject has a new systemic steroid therapy
* Subject is unlikely to comply with the procedures scheduled in the protocol
* Subject has a known allergic reaction to the medication
* Subject is pregnant or breastfeeding
* Patient participates in another clinical trial within 30 days prior to study entry or 30 days after end of the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Variations in the Sino-nasal-outcome test SNOT-20 adapt CF (primary nasal parameters: obstruction of nasal breathing, sneeze stimulus, permanent nose running, thick-mucous nasal discharge, earaches) | day 1, 29, 57 and 85

SECONDARY OUTCOMES:
Variations in the Sino-nasal-outcome test SNOT-20 adapt CF (secondary nasal parameters, general quality of live parameters and total SNOT 20 adapt. CF score) | day 1, 29, 57 and 85
Changes of pathological alterations visible in MRT images of nose and paranasal sinuses (in selected patients) | day 1, 29, 57, 85
Changes in the nasal lavage fluid and in the serological markers of inflammation | day 1, 29, 57 and 85
Changes in rhinoscopic findings | day 1, 29, 57 and 85
Changes in rhinomanometric findings | day 1, 29, 27 and 85
Incidence of rhinosinusitic and pulmonary exacerbations during therapy | day 1 - 85
Need for decongestants or nasal lavage during treatment | day 1 - 85

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Mainz, M.D., Study Chair — University of Jena
Locations (2):
- Germany (2):
  - Universitäts-Kinderklinik, Tübingen, Baden-Würtemberg
  - Mukoviszidosezentrum der Friedrich-Schiller-Universität, Jena, Thuringia

REFERENCES:
- [Background] Mainz JG, Michl R, Arnold C. Response to Karadag. J Cyst Fibros. 2014 Sep;13(5):602-3. doi: 10.1016/j.jcf.2014.07.005. Epub 2014 Jul 28. No abstract available. PMID 25081561
- [Result] Mainz JG, Schien C, Schiller I, Schadlich K, Koitschev A, Koitschev C, Riethmuller J, Graepler-Mainka U, Wiedemann B, Beck JF. Sinonasal inhalation of dornase alfa administered by vibrating aerosol to cystic fibrosis patients: a double-blind placebo-controlled cross-over trial. J Cyst Fibros. 2014 Jul;13(4):461-70. doi: 10.1016/j.jcf.2014.02.005. Epub 2014 Mar 1. PMID 24594542